CLINICAL TRIAL: NCT00614484
Title: Phase I/II Study of Combined Chemotherapy and High Dose, Accelerated Proton Radiation for the Treatment of Locally Advanced Non-Small Cell Lung Carcinoma
Brief Title: Chemotherapy and Proton Radiation for the Treatment of Locally Advanced Lung Cancer
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Low participant enrollment rates. Significant comparative data not obtained.
Sponsor: Loma Linda University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OSR #49168
Record Dates: First submitted 2007-12-26; First posted 2008-02-13 (Estimated); Results first posted 2014-05-22 (Estimated); Last update posted 2014-05-22 (Estimated); Status verified 2014-04

CONDITIONS: Locally Advanced Non-Small Cell Lung Cancer
Keywords: Proton; Radiation
MeSH Terms: interventions — Protons; Paclitaxel; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Proton therapy with chemotherapy (Experimental): Induction Chemotherapy - Two cycles Taxol 200mg/m2 and Carboplatin AUC6 on day 1 and day 22. Weekly chemotherapy concurrent with radiotherapy Taxol 50mg/m2 and Carboplatin AUC 2 weekly for 5 weeks.
  Proton therapy - 76 Gy in 5 weeks to lung tumor.
  Interventions: Radiation: Proton Radiation Therapy; Drug: Taxol; Drug: Carboplatin

INTERVENTIONS:
Radiation: Proton Radiation Therapy — A five week coarse of proton radiotherapy begins on day 28 and is given once daily for the first two weeks and twice daily for the final 3 weeks. The total dose given with proton beam is 76 Gy. Weekly chemotherapy with carboplatin and taxol is given during proton therapy.
Drug: Taxol — 200 mg/m2, IV, for 2 cycles followed by 50 mg/m2 weekly for 5 weeks during radiotherapy.
  Other Names: Paclitaxel
Drug: Carboplatin — AUC 6, IV, for two cycles followed by AUC 2 weekly for 5 weeks during radiotherapy.

SUMMARY:
The purpose of this study is to determine the effectiveness of proton beam radiotherapy combined with chemotherapy for treatment of locally advanced non-small cell lung cancer.

ELIGIBILITY:
Inclusion Criteria:

* Clinical stage 2, 3A or 3B (unresectable)
* Histologic evidence of non-small cell carcinoma
* Age > 18 years
* Karnofsky performance status 70 or greater
* No prior radiation to the chest
* No previous chemotherapy

Exclusion Criteria:

* Clinical stage 1 or 4
* Previous malignancies except for non-melanoma skin cancer unless disease free for > 3 years

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 1999-08; Primary Completion 2011-06 (Actual); Study Completion 2011-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A. Bush, MD, Principal Investigator — Loma Linda University Department of Radiation Medicine; Jerry D. Slater, MD, Study Chair — Loma Linda University Department of Radiation Medicine
Locations (1):
- Loma Linda University Medical Center, Loma Linda, California, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subject were recruited from the radiation oncology clinic from 11/99 through 4/11.
Groups:
- Treatment With Chemotherapy and Proton Beam Radiotherapy.: Induction chemotherapy with two cycles of taxol and carboplatin given on day 1 and day 15. A five week coarse of proton radiotherapy begins on day 28 and is given once daily for the first two weeks and twice daily for the final 3 weeks. Weekly chemotherapy with carboplatin and taxol is given during proton therapy.
Period: Overall Study
Arm/Group | Treatment With Chemotherapy and Proton Beam Radiotherapy.
Started | 28
Completed | 28
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: 28 subjects were enrolled and received the study treatment. All 28 were followed for treatment outcomes.
Arm/Group | Treatment With Chemotherapy and Proton Beam Radiotherapy.
Number analyzed (Participants) | 28
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 13
  >=65 years | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 66 (8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 17
Region of Enrollment [Number; unit: participants]
  United States | 28

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival.
Description: Median survival time following treatment.
Time Frame: Monthly for duration of participant lifespan. Average lifespan 1-2 years
Measure: Median (95% Confidence Interval); unit: Months
Groups:
- Chemothrapy and Proton Therapy: Induction chemotherapy with two cycles of taxol and carboplatin given on day 1 and day 15. A five week coarse of proton radiotherapy begins on day 28 and is given once daily for the first two weeks and twice daily for the final 3 weeks. Weekly chemotherapy with carboplatin and taxol is given during proton therapy.
Arm/Group | Chemothrapy and Proton Therapy
Number analyzed (Participants) | 28
Months | 15 [10 to 20]

2. Secondary Outcome: Treatment Related Toxicities.
Description: grade 3 or higher esophageal toxicity
  Toxicity is categorized either early or late phase.
  Early phase- toxicity occurring during or within 30 days s/p treatment Late phase- toxicity occurring thereafter
Time Frame: Monthly for duration of participant lifespan. Average lifespan 1-2 years
Measure: Number; unit: participants
Groups:
- Chemotherapy and Proton Therapy: Induction chemotherapy with two cycles of taxol and carboplatin given on day 1 and day 15. A five week coarse of proton radiotherapy begins on day 28 and is given once daily for the first two weeks and twice daily for the final 3 weeks. Weekly chemotherapy with carboplatin and taxol is given during proton therapy.
Arm/Group | Chemotherapy and Proton Therapy
Number analyzed (Participants) | 28
participants | 2

ADVERSE EVENTS:
Time Frame: Participants were followed for the duration of their lifespan, an average of 1-2 years
Arm/Group | Treatment With Chemotherapy and Proton Beam Radiotherapy.
Serious Adverse Events (participants affected / at risk) | 4/28
Other Adverse Events (participants affected / at risk) | 12/28
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With Chemotherapy and Proton Beam Radiotherapy. (N=28)
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 2 (2) — Grade 3 pneumonitis
Pulmonary hemorrage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Esophageal Fistula (Respiratory, thoracic and mediastinal disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With Chemotherapy and Proton Beam Radiotherapy. (N=28)
Esophagitis (Respiratory, thoracic and mediastinal disorders) | 12 (12) — Grade 1/2 esophagitis

LIMITATIONS AND CAVEATS:
Slow enrollment over a long time period limits the conclusions that can be drawn.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes